CLINICAL TRIAL: NCT02853123
Title: A Randomised, Double-blind, Cross-over Study to Evaluate the Effect of 6 Weeks Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (5/5 µg) Compared With Tiotropium (5 µg), Both Delivered by the Respimat® Inhaler, on Breathlessness During the Three Minute Constant Speed Shuttle Test (3min CSST) in Patients With Chronic Obstructive Pulmonary Disease (COPD). [OTIVATO TM]
Brief Title: Effect of Tiotropium + Olodaterol on Breathlessness in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.28; 2015-002974-20 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tiotropium + Olodaterol (Experimental): Patients will receive tiotropium 5mcg + olodaterol 5mcg in a fixed dose combination once daily.
  Interventions: Drug: Tiotropium; Drug: Olodaterol
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — fixed dose combination once daily
  Arms: Tiotropium + Olodaterol
Drug: Olodaterol — fixed dose combination once daily
  Arms: Tiotropium + Olodaterol
Drug: Tiotropium
  Arms: Tiotropium

SUMMARY:
The primary objective of the present study is to evaluate the effect of tiotropium + olodaterol fixed dose combination (FDC) compared to tiotropium monotherapy on the intensity of breathlessness during the 3min constant speed shuttle test (CSST).

A secondary objective is to explore the relationship between reductions in breathlessness during the 3min CSST and reductions in breathlessness during activities of everyday living as measured by the dyspnea domain of the Chronic Respiratory Questionnaire (CRQ) following bronchodilator therapy.

ELIGIBILITY:
Inclusion criteria:

* Patients must sign an informed consent consistent with International Conference on Harmonization Good Clinical Practice guidelines prior to participation in the trial, including medication washout and restrictions
* Diagnosis of Chronic Obstructive Pulmonary Disease and relatively stable airway obstruction: post bronchodilator 30%<= Forced Expiratory Volume in 1st second (FEV1)<80% of predicted normal (European Coal and Steel Community) and a post bronchodilator FEV1/Forced Vital Capacity<0.70 at visit 1
* Male or female patients >=40 and =<75 years of age on day of signing consent.
* Current or ex-smokers with a smoking history > 10 pack-years. Patients who have never smoked cigarettes must be excluded.
* Baseline Dyspnea Index score< 8 at visit 0.
* Hyperinflation at rest, defined as Functional Residual Capacity > 120% predicted at visit 1.
* Borg dyspnea score >=4 at the end of 3min Constant Speed Shuttle Test at visit 2
* Perform technically acceptable pulmonary function tests (spirometry and body plethysmography) and complete multiple shuttle tests during the study period
* Inhale medication in a competent manner from the Respimat® inhaler and from a metered dose inhaler

Exclusion criteria:

* Significant disease other than Chronic Obstructive Pulmonary Disease (COPD); a significant disease which, in the investigator's opinion, may (i) put the patient at risk (ii) influence the study results or (iii) cause concern regarding the patient's ability to participate
* Clinically relevant abnormal baseline haematology, blood chemistry, in the investigator's opinion, or creatinine >x2 Upper Limit Normal will be excluded regardless of clinical condition
* Current documented diagnosis of asthma
* COPD exacerbation in the 6 weeks prior to screening
* Diagnosis of thyrotoxicosis
* History of myocardial infarction within 6 months of screening
* Life-threatening cardiac arrhythmia (investigator judgment)
* Known active tuberculosis
* Any malignancy unless free of disease for at least 5 years (treated basal cell carcinoma or squamous cell skin cancers are allowed)
* History of cystic fibrosis
* Clinically relevant bronchiectasis (investigator judgment)
* Severe emphysema requiring endobronchial interventions within 6 months prior to screening
* History of significant alcohol or drug abuse (investigator judgment)
* Any contraindications for exercise testing
* Patients who have undergone thoracotomy with pulmonary resection
* Treatment with any oral or patch ß-adrenergics
* Treatment with oral corticosteroid medication at unstable doses or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Treatment with antibiotics for any reason within 4 weeks of screening
* Patients being treated with Phosphodiesterase Type 4 (PDE4) inhibitors within 3 months of screening visit should not be enrolled and PDE4 inhibitors should not be withdrawn for the purpose of enrolling in this study
* Regular use of daytime oxygen therapy for >1 hour per day and in the investigator's opinion will be unable to abstain from use during clinic visits
* Completion of a pulmonary rehabilitation program 6 weeks prior to screening or currently in a program
* Limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea, such as arthritis in the leg, angina pectoris, claudication, morbid obesity
* Endurance time >=12 minutes during the incremental shuttle walk test
* Oxygen saturation < 85% (on room air) at rest or during exercise.
* Taken an investigational drug within 1 month or 6 half-lives or in case the investigational drug class is listed within the washout period specified prior to screening visit
* Known hypersensitivity to ß-adrenergics and/or anticholinergic drugs, Benzalkonium Chloride, Ethylenediaminetetraacetic acid or any other component of the Respimat® inhalation solution
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Women of childbearing potential not using a highly effective method of birth control
* Previously been randomized in this study or are currently participating in another study
* Unable to comply with pulmonary medication restrictions prior to randomization

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (13):
- Belgium (3):
  - Genk - PRAC Janssens, E., Genk
  - Hasselt - PRAC Aumann, J-L, Hasselt
  - UZ Leuven, Leuven
- Canada (4):
  - McMaster Univ. Medical Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - IUCPQ (Laval University), Québec
- Germany (3):
  - Klinische Forschung Berlin GbR, Berlin
  - IKF Pneumologie GmbH & Co. KG, Frankfurt am Main
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Zuyderland Medisch Centrum, Heerlen
  - Gelre Ziekenhuis Zutphen, Zutphen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, active-controlled, 2-period crossover, Phase IV study to evaluate the effects of once daily administration of orally inhaled tiotropium + olodaterol fixed dose combination compared with tiotropium on the intensity of breathlessness in patients with Chronic Obstructive Pulmonary Disease (COPD).
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which then ensured that all patients met all inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any specific entry criteria were violated.
Groups:
- (Tiotropium 5 Microgram (μg))/(Tiotropium + Olodaterol 5/5 μg): Patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium (Tio) inhalation solution (2.5 μg per actuation) once a day, in the morning for a period of 6 weeks in period 1 followed by a 3 week washout period. In period 2, patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium + Olodaterol (Tio+Olo) fixed dose combination (FDC) inhalation solution (2.5/2.5 μg per actuation) once a day, in the morning for a period of 6 weeks.
- (Tiotropium + Olodaterol 5/5 μg)/(Tiotropium 5 μg): Patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium + Olodaterol (Tio+Olo) fixed dose combination (FDC) inhalation solution (2.5/2.5 μg per actuation) once a day, in the morning for a period of 6 weeks in period 1 followed by a 3 week washout period. In period 2, patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium (Tio) inhalation solution (2.5 μg per actuation) once a day, in the morning for a period of 6 weeks.
Period: Treatment Period 1
Arm/Group | (Tiotropium 5 Microgram (μg))/(Tiotropium + Olodaterol 5/5 μg) | (Tiotropium + Olodaterol 5/5 μg)/(Tiotropium 5 μg)
Started | 52 | 54
Completed | 52 | 51
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 3
Period: Washout Period
Arm/Group | (Tiotropium 5 Microgram (μg))/(Tiotropium + Olodaterol 5/5 μg) | (Tiotropium + Olodaterol 5/5 μg)/(Tiotropium 5 μg)
Started | 52 | 51
Completed | 51 | 48
Not Completed | 1 | 3
Not completed — Worsening of COPD | 0 | 3
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2
Arm/Group | (Tiotropium 5 Microgram (μg))/(Tiotropium + Olodaterol 5/5 μg) | (Tiotropium + Olodaterol 5/5 μg)/(Tiotropium 5 μg)
Started | 51 | 48
Completed | 51 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set was nested within the randomized set (RS) and included all patients who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Total Subjects: This patient set was nested within the randomized set (RS) and included all patients who were dispensed study medication and were documented to have taken any dose of study medication.
Arm/Group | Total Subjects
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] — The age data are presented by years. Population: TS
  Years | 63.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — The sex data are presented by count of participants. Population: TS
  Participants
    Female | 40
    Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race data are presented by count of participants. Ethnicity was not captured in this trial. Population: TS
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 105
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intensity of Breathlessness Measured Using the Modified Borg Scale at the End of the 3 Minute (Min) Constant Speed Shuttle Test After 6 Weeks of Treatment.
Description: At 3 min or end of exercise (if 3 min not achieved), patients were asked to estimate the intensity of breathing discomfort that they were experiencing by matching their subjective estimate to descriptive phrases that best described the intensity of each sensation using the Modified Borg Scale (MBS-S). The modified Borg scale is 10-point subjective scoring system, in which a patient rates effort of exertion while performing a particular activity. The scale is 0 to 10, the higher the score, the greater the perceived difficulty. Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: Full analysis set (FAS): This patient set was nested within the treated set (TS) and included patients who had baseline measurement and at least one post-baseline measurement for the primary endpoint. FAS including participants with available data for change from baseline in intensity of breathlessness after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Groups:
- Tiotropium 5 Microgram (μg): Patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium (Tio) inhalation solution (2.5 μg per actuation) once a day, in the morning for a period of 6 weeks.
- Tiotropium + Olodaterol 5/5 μg: Patients inhaled 2 puffs from the Respimat® Inhaler of the Tiotropium + Olodaterol (Tio+Olo) fixed dose combination (FDC) inhalation solution (2.5/2.5 μg per actuation) once a day, in the morning for a period of 6 weeks.
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 100 | 101
Unit on Scale | -0.968 (0.137) | -1.325 (0.136)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; The adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p = 0.0217, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = -0.357, 95% CI 2-sided [-0.661 to -0.053], Standard Error of Mean 0.153 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

2. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for Inspiratory Capacity Measured Prior to Exercise
Description: Inspiratory Capacity (IC) is a standard measurement for the assessment of lung function. IC measurements were performed prior to the 3min Constant Speed Shuttle Test (CSST) (at rest). Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for inspiratory capacity measured prior to exercise after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 100 | 101
Litre (L) | 0.279 (0.040) | 0.464 (0.039)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; IC measured prior to exercise, the adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p < .0001, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = 0.185, 95% CI 2-sided [0.106 to 0.265], Standard Error of Mean 0.040 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

3. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for Inspiratory Capacity Measured at the End of Exercise
Description: Inspiratory Capacity (IC) is a standard measurement for the assessment of lung function. IC measurements were performed at the end of the 3min Constant Speed Shuttle Test (CSST). Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for inspiratory capacity measured end of exercise after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 98 | 100
Litre (L) | 0.256 (0.034) | 0.322 (0.034)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; IC measured end of exercise, the adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p = 0.0852, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.009 to 0.141], Standard Error of Mean 0.038 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

4. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for 1 Hour Post-dose Forced Expiratory Volume
Description: Forced Expiratory Volume in 1st second (FEV1) is a standard measurement for the assessment of lung function. The best of 3 efforts was defined as the highest FEV1, each obtained on any of 3 manoeuvres meeting the American Thoracic Society (ATS) criteria (to a maximum of 5 attempts). Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for FEV1 after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 99 | 103
Litre (L) | 0.163 (0.021) | 0.318 (0.021)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = 0.155, 95% CI 2-sided [0.117 to 0.194], Standard Error of Mean 0.020 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

5. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for 1 Hour Post-dose Forced Vital Capacity
Description: Forced Vital Capacity (FVC) is a standard measurement for the assessment of lung function. The best of 3 efforts was defined as the highest FVC, each obtained on any of 3 manoeuvres meeting the American Thoracic Society (ATS) criteria (to a maximum of 5 attempts). Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for FVC after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 99 | 103
Litre (L) | 0.258 (0.040) | 0.459 (0.039)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .0001, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = 0.201, 95% CI 2-sided [0.134 to 0.267], Standard Error of Mean 0.034 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

6. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for Intensity of Breathlessness (MBS-S) at 1, 2 and 2.5 Minute (Min) During the 3 Min Constant Speed Shuttle Test
Description: At 1, 2 and 2.5 min during exercise, patients were asked to estimate the intensity of breathing discomfort that they were experiencing by matching their subjective estimate to descriptive phrases that best described the intensity of each sensation using the Modified Borg Scale (MBS-S). At 3 min or end of exercise (if 3 min not achieved), patients were asked to estimate the intensity of breathing discomfort that they were experiencing by matching their subjective estimate to descriptive phrases that best described the intensity of each sensation using the Modified Borg Scale (MBS-S). The modified Borg scale is 10-point subjective scoring system, in which a patient rates effort of exertion while performing a particular activity. The scale is 0 to 10, the higher the score, the greater the perceived difficulty. Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for MBS-S after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 100 | 101
Unit on Scale
  1 min | -0.685 (0.081) | -0.793 (0.081)
  2 min | -0.839 (0.102) | -1.079 (0.101)
  2.5 min | -0.846 (0.127) | -1.164 (0.126)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; 1 min, the adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p = 0.2645, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = -0.108, 95% CI 2-sided [-0.300 to 0.083], Standard Error of Mean 0.096 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)
Statistical Analysis 2: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; 2 min, the adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p = 0.0267, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = -0.240, 95% CI 2-sided [-0.452 to -0.028], Standard Error of Mean 0.107 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)
Statistical Analysis 3: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; 2.5 min, the adjusted means (SE) are obtained from fitting an Mixed-effects Model Repeated Measures (MMRM) model including treatment and period as fixed effects, patient as a random effect, and period baseline and patient baseline as covariates, compound symmetry covariance structure for within-patient variation; Test type: Superiority; p = 0.0258, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = -0.318, 95% CI 2-sided [-0.596 to -0.039], Standard Error of Mean 0.140 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

7. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for Chronic Respiratory Questionnaire - Self Administered Individualized (CRQ-SAI) Dyspnoea Domain Score
Description: CRQ-SAI refers to the CRQ-Self-administered individualized format as it contains a dyspnea domain that is individualized to each patient. This version was derived from the original CRQ tool & therefore, is scored on 7-point Likert-type scale (1: maximum impairment to 7: no impairment) for each 4 domains covering: dyspnea, fatigue, emotional function & mastery. Dyspnea items may be selected from list of 26 suggested items or written in by the patients. The patients are asked to select up to 5 activities associated with breathlessness that they perform frequently and are most important to them. The scores for each question of each domain were added together and divided by the number of questions answered in each domain. The higher scores indicate better health-related quality of life in the respective domain. Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for CRQ-SAI questionnaire after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 93 | 96
Unit on Scale | 0.640 (0.091) | 0.610 (0.089)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8025, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.268 to 0.208], Standard Error of Mean 0.120 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

8. Secondary Outcome: Change From Baseline After 6 Weeks of Treatment for Chronic Respiratory Questionnaire - Self Administered Standardized (CRQ-SAS) Dyspnoea Domain Score
Description: CRQ-SAS was questionnaire to assess patients' perception of COPD and measures the impact of COPD on their life. This version was derived from the original CRQ tool & therefore, is scored on 7-point Likert-type scale (1: maximum impairment to 7: no impairment) for each 4 domains covering: dyspnea, fatigue, emotional function & mastery. The CRQ-SAS refers to the CRQ-Self-administered standardized format & contains 20 questions. The first part of the questionnaire contains 5 standardized dyspnea questions and the patients must indicate how much shortness of breath they have experienced while performing each of these 5 activities. The scores for each question of each domain were added together and divided by the number of questions answered in each domain. The higher scores indicate better health-related quality of life in the respective domain. Measure type is actually Adjusted Mean Change from Baseline.
Time Frame: Baseline and week 6
Population: FAS including participants with available data for change from baseline for CRQ-SAS questionnaire after 6 weeks of treatment.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg
Number analyzed (Participants) | 100 | 102
Unit on Scale | 0.325 (0.088) | 0.415 (0.087)
Statistical Analysis 1: Comparison: Tiotropium 5 Microgram (μg) vs Tiotropium + Olodaterol 5/5 μg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3634, Mixed Effect Model Repeated Measures; Kenward-Roger approximation of denominator was used for degrees of freedom; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.106 to 0.286], Standard Error of Mean 0.099 — Mean difference means the treatment difference vs. Tiotropium (i.e. Tiotropium/Olodaterol - Tiotropium)

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after last drug administration, up to 18 weeks.
Description: Treated set (TS) (This patient set was nested within the Randomised set (RS) and included all patients who were dispensed study medication and were documented to have taken any dose of study medication.) was used for patient safety analyses.
Arm/Group | Tiotropium 5 Microgram (μg) | Tiotropium + Olodaterol 5/5 μg | Total Subjects
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 1/100 | 5/105 | 6/106
Other Adverse Events (participants affected / at risk) | 21/100 | 31/105 | 44/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 Microgram (μg) (N=100) | Tiotropium + Olodaterol 5/5 μg (N=105) | Total Subjects (N=106)
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium 5 Microgram (μg) (N=100) | Tiotropium + Olodaterol 5/5 μg (N=105) | Total Subjects (N=106)
Viral upper respiratory tract infection (Infections and infestations) | 13 | 14 | 23
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT02853123/SAP_000.pdf
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT02853123/Prot_001.pdf